CLINICAL TRIAL: NCT01104714
Title: Pharmacogenetic and Pharmacokinetic Aspects of the Response to Chemotherapy Induction Using Docetaxel, Cisplatin and 5-Fluorouracile (TPF)in ORL Cancers
Brief Title: Pharmacogenetic Response to Chemotherapy Induction for ORL Cancers
Acronym: APPROCHE ORL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2008/BL-01; 2008-006874-14 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma, Squamous Cell; Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms
MeSH Terms: conditions — Carcinoma, Squamous Cell; Mouth Neoplasms; Oropharyngeal Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Surplus blood, tumor tissue from biopsies, and DNA will be stocked in the Biothèque of the Nîmes University Hospital
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: As the trial progresses, patients will be classified as either chemotherapy responders or non-responders.

SUMMARY:
The purpose of this study is to determine if there is a correlation between tumor response after 3 doses of chemotherapy by induction using Docetaxel, Cisplatine and 5-Fluorouracile for advanced stage epidermoid carcinomas of the upper aero digestive tract and the presence of one or a combination of 3 genetic polymorphisms and/or 5 intra-tumoral transcriptional modifications.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma originating in the mouth, oropharynx, larynx or hypopharynx has been histologically documented.
* The disease is at one of the following UICC 2002 stages, regardless of ganglion status: T3 MO or T4 MO
* Treatment via chemotherapy, radiotherapy or surgery (except for the diagnostic biopsy) has not started
* The pluridisciplinary committee as ruled out surgical options for technical or functional reasons
* Absence of distant metastases
* OMS general health status between 0 and 2
* Patient has given informed consent
* Patient is affiliated with a social security system

Exclusion Criteria:

* Undifferentiated squamous cell carcinomas in the nasopharynx (UCNT)
* Another cancer priorly treated with one of the following chemotherapies: Docetaxel, Cisplatin, 5-Fluorouracile
* Creatininemia > 2 mg/dl and/or creatinine clearance < 60ml/min
* Patient under guardianship
* Presence of another severe pathology including:

  * severe or chronic cardiac, renal and/or hepatic insufficiencies
  * severe medullary hypoplasia
  * severe autoimmune disease
  * psychosis or senility

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study have been diagnosed with an advanced stage squamous cell carcinoma in the buccal, oropharyngeal, laryngeal or hypopharyngeal areas.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
%change in tumor volume before and after chemotherapy (baseline versus 62 days) | 62 days
  Tumor volume is calculated according to Labadie et al 2000

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lallemant, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (14):
- France (14):
  - CH d'Alès, Alès
  - CHU de Bordeaux - Groupe Hospitalier Saint-André, Bordeaux
  - CHU de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU de Grenoble, Grenoble
  - Centre de Lutte Contre le Cancer - Centre Oscar Lambret, Lille
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Val d'Aurelle - Paul Lamarque, Montpellier
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Centre de Lutte Contre le Cancer - Institut Claudius Regaud, Toulouse
  - Pharmacologie Clinique, expérim. des anticancéreux, CLCC Claudius Regaud, Toulouse
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse
  - CHRU de Toulouse - Hôpital Larrey, Toulouse
  - CHRU de Toulouse - Hôpital Purpan, Toulouse

REFERENCES:
- [Background] Labadie RF, Yarbrough WG, Weissler MC, Pillsbury HC, Mukherji SK. Nodal volume reduction after concurrent chemo- and radiotherapy: correlation between initial CT and histopathologic findings. AJNR Am J Neuroradiol. 2000 Feb;21(2):310-4. PMID 10696014